CLINICAL TRIAL: NCT02591823
Title: Observational Study of Hair Fall in Rheumatoid Arthritis Patients Treated With Low Dose Methotrexate
Brief Title: Hair Fall in Patients on Low Dose Methotrexate
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Columbia Asia (Other)
Responsible Party: Principal Investigator, Dr.Sharath Kumar, Consultant Rheumatologist, Columbia Asia
Other Study IDs: IEC/2015/RP/18
Record Dates: First submitted 2015-10-28; First posted 2015-10-30 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Alopecia; Rheumatoid Arthritis; Methotrexate Adverse Reaction
MeSH Terms: conditions — Alopecia; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Healthy Controls: Healthy subject who accompanying patients to rheumatology OPD or healthy subjects who are staff at Columbia Asia Hospital,Bangalore.
- Cases (patients on methotrexate): Subjects attending the rheumatology OPD of Columbia Asia hospitals bengaluru, who are diagnosed as having Rheumatoid arthritis and fulfill the ACR/ EULAR 2010 classification criteria for rheumatoid arthritis and are started on low dose methotrexate will included as cases

SUMMARY:
Low dose methotrexate used in rheumatoid arthritis is considered very safe and has a side effect profile very different from that seen with high dose methotrexate used in oncology. Hair fall has been found to occur in high dose methotrexate but there is no data regarding the same when methotrexate is used in low dose.Thus this observational case control study is being undertaken to determine whether rheumatoid arthritis patients really need to be concerned about hair fall when on low dose methotrexate.

ELIGIBILITY:
Inclusion Criteria:

For Cases

* Subjects should be above 18 years of age.
* Diagnosed with rheumatoid arthritis and fulfilling the ACR EULAR 2010 criteria.
* Should be initiated on methotrexate
* Willing to follow up

For Controls

-Subjects should be above 18 years of age.

Exclusion Criteria:

For Cases

* Subjects with prior exposure to methotrexate in the last 6 months
* Subjects suffering from Thyroid (hypothyroidism)
* Subjects on leflunomide, or having received leflunomide in the last 6 months
* Subjects currently on cyclophosphamide or having received cyclophosphamide in the last 3 months.
* Subjects on psychiatric treatment or depression illness.
* Subjects who have overlap with other rheumatological disorders which can cause hair fall.
* Subjects in 1-5 months of post-partum or post-natal period.
* Subjects with female pattern baldness
* Subjects with androgenetic alopecia
* Subjects with alopecia aereta
* Subjects with other scalp conditions which can predispose to hair fall

For Controls

* Subjects having any family history of alopecia.
* Subjects suffering from thyroid.
* Subjects having any history of anemia.
* Subjects under 1-5 months of post-partum or post-natal period.
* Subjects on medications which can cause hair fall.
* Subjects on methotrexate for other reasons.
* Subjects with female pattern baldness
* Subjects with androgenetic alopecia
* Subjects with alopecia aereta
* Subjects with other scalp conditions which can predispose to hair fall

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cases will consist of consecutive patients diagnosed with rheumatoid arhtiritis in the rheumatology OPD of Columbia Asia hospitals,Bengaluru who are started on methotrexate.
  Control population will consist of healthy volunteers (relatives of patients attending the rheumatology OPD or staff in the hospital)
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-04 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Mean change in number of hair strands obtained by the hair pull test at the baseline and at 3 weeks among RA patients on methotrexate in comparison to the mean change in the same number among controls. | 3 weeks
  Mean change in number of hair strands obtained by the hair pull test at the start of the trial and at 3 weeks among rheumatoid arthritis patients on methotrexate in comparison to the mean change in the same number among health controls

SECONDARY OUTCOMES:
Mean change in number of hair strands obtained by the hair pull test at baseline and at 2 months among RA patients on methotrexate in comparison with mean change in the same number among controls. | 2 months
Mean change in number of hair strands obtained by the hair pull test at the start of the trial and at 3 months among RA patients on methotrexate in comparison to the mean change in the same number among control. | 3 Months
Mean difference in number of subjects having an abnormal hair pull test (defined as > 5 hairs) at baseline and at 3 weeks in patients with RA on methotrexate and compare the same with the mean difference. | 3 weeks
Mean difference in number of subjects having an abnormal hair pull test at baseline and at 2 months in patients with RA patients on methotrexate and compare the same with the mean difference. | 2 months
Mean difference in number of subjects having an abnormal hair pull test at baseline and at 3 months in patients with RA patients on methotrexate and compare the same with the mean difference. | 3 months
Difference in number of subjects having an anagen hair among the the hair obtained by hair pull test (normal = 0) at 3 weeks between RA patients on methotrexate and controls. | 3 weeks
Difference in number of subjects having an anagen hair among the hair obtained by hair pull test (normal = 0) at 2 months between RA patients on methotrexate and controls. | 2 months
Difference in number of subjects having an anagen hair among the the hair obtained by hair pull test (normal = 0) at 3 months between rheumatoid arthritis patients on methotrexate and healthy controls. | 3 Months
Difference in the mean number of hair obtained at the time of inclusion in the study among rheumatoid arthritis patients and health controls | 0 month
Determine the difference in number of subjects having an abnormal hair pull test at baseline in patients with RA patients on methotrexate and controls. | 0 month
Determine the difference in number of subjects having an anagen hair among the the hair obtained by hair pull test (normal = 0) at inclusion in the study between RA patients on methotrexate and healthy controls. | 0 month

CONTACTS AND LOCATIONS:
Overall Officials: Sharath Kumar, MBBS,MD,DNB, Principal Investigator — Columbia Asia Hospitals,Bangalore
Locations (1):
- Columbia Asia Hospitals, Bangalore, Karnataka, India

REFERENCES:
- [Background] Malaviya AN, Sharma A, Agarwal D, Kapoor S, Garg S, Sawhney S. Low-dose and high-dose methotrexate are two different drugs in practical terms. Int J Rheum Dis. 2010 Oct;13(4):288-93. doi: 10.1111/j.1756-185X.2010.01564.x. Epub 2010 Aug 16. PMID 21199463
- [Background] Emery P, Breedveld FC, Lemmel EM, Kaltwasser JP, Dawes PT, Gomor B, Van Den Bosch F, Nordstrom D, Bjorneboe O, Dahl R, Horslev-Petersen K, Rodriguez De La Serna A, Molloy M, Tikly M, Oed C, Rosenburg R, Loew-Friedrich I. A comparison of the efficacy and safety of leflunomide and methotrexate for the treatment of rheumatoid arthritis. Rheumatology (Oxford). 2000 Jun;39(6):655-65. doi: 10.1093/rheumatology/39.6.655. PMID 10888712
- [Background] Hansen HH, Selawry OS, Holland JF, McCall CB. The variability of individual tolerance to methotrexate in cancer patients. Br J Cancer. 1971 Jun;25(2):298-305. doi: 10.1038/bjc.1971.38. PMID 4256007